CLINICAL TRIAL: NCT02011035
Title: Evaluating the Clinical Efficacy and Safety of Colfelx
Brief Title: Evaluating the Clinical Efficacy and Safety of Colflex
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Peter Jones, Director of the Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Other Study IDs: B2013:133
Record Dates: First submitted 2013-09-30; First posted 2013-12-13 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Personal Satisfaction
Keywords: Oral health; Mouth health; Halitosis; Oral bacteria; Sore throat; Colds
MeSH Terms: conditions — Personal Satisfaction; Halitosis; Pharyngitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to test the safety and efficacy of Colflex, an oral spray created by Innotech Nutrition, on human subjects to measure changes on frequency/duration of colds and sore throats, as well as dental and oral health changes.

ELIGIBILITY:
Inclusion Criteria:

* availability to give written consent
* age 18-60, men and women (who are not pregnant or nursing)
* people in good health
* able to follow protocol
* must be experiencing a sore throat or cold at least once a year

Exclusion Criteria:

* smokers
* liver and kidney disease
* inflammatory bowel disease
* pancreatitis
* gallbladder or biliary disease
* neurolgical/psychological disease
* bleeding disorders
* platelet abnormatilies
* gastrointestinal disorders that could interfere with fat absorption
* serum triglycerides > 500 mg/dL and/or total cholesterol > 300 mg/dL
* hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure > 100 Hg
* BMI >30
* consume or planned to consume anticoagulant, hypertension, or lipid lowering medications
* reported consumption of more than 2 alcoholic drinks/day or history of alcoholism or drug dependence
* reported use of experimental medication within 1 month prior to the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents in town
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of colds/sore throats | 30 days
  Using a self-reported scale to assess the frequency and during of colds and sore throats at screening, and at baseline and endpoint of treatments

SECONDARY OUTCOMES:
Assessment of oral pathogenic bacteria | 30 days
  A mouth swab will be taken to measure pathogenic bacteria (Straph, Strep), and a mouth swab will be used for the BANA test to test for periodontal disease causing bacteria.

OTHER OUTCOMES:
Effect on plasma lipid profile and enzyme measurements | 30 days
  Exploratory efficacy measures include lipid profile, (TC, HDL, TG), and liver enzymes
Measurement of oral halitosis | 30 days
  A breath sample is taken to measure volatile sulphur compounds using a halimeter.

CONTACTS AND LOCATIONS:
Locations (1):
- RCFFN: University of Manitoba, Winnipeg, Manitoba, Canada